CLINICAL TRIAL: NCT06881706
Title: Relationship Between Biochemical and Anthropometric Variables and CD36 Levels in Metabolic Syndrome Patients After Low Calorie Diet
Brief Title: Link Between Biochemical, Anthropometric Variables and CD36 in Metabolic Syndrome After a Low-calorie Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Duygu MATARACI DEĞİRMENCİ, Assistant Professor, Ordu University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Metabolic syndrome and CD36
Record Dates: First submitted 2025-02-25; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Metabolic Syndrome; Weight Loss
Keywords: metabolic syndrome; weight loss; cd36; fatty acids; fatty acid receptor
MeSH Terms: conditions — Metabolic Syndrome; Weight Loss | interventions — Nutrition Therapy

STUDY DESIGN:
Intervention Model Description: There are 2 groups in the study. Both groups consist of individuals with newly diagnosed metabolic syndrome. The first group (intervention group) is the group that applied a weight loss diet and achieved weight loss. The second group (control group) is the group that did not apply a diet and did not achieve weight loss.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): At the beginning of the study, all participants were given a hypocaloric diet to induce weight loss. Individuals who followed the diet and lost at least 5% of their starting weight constituted this group.
  Interventions: Other: medical nutrition therapy
- Control Group (No Intervention): At the beginning of the study, all participants were given a hypocaloric diet to induce weight loss. Individuals who did not follow the diet and did not lose at least 5% of their starting weight constituted this group.

INTERVENTIONS:
Other: medical nutrition therapy — Medical nutrition treatment was planned for all participants with metabolic syndrome. A diet plan was created considering age, gender, blood findings and nutritional habits. Individuals with MetS were given a weight loss diet planned at the basal energy level calculated with the Harris-Benedict equation and applied for 8 weeks. Individuals who applied the weight loss diet were targeted to lose at least 5% of their initial weight at the end of 8 weeks. Individuals who strictly followed the given medical nutrition treatment and achieved the targeted weight loss formed the intervention group, and individuals who did not follow the medical nutrition treatment formed the control group. At the end of the 8 weeks, all parameters, blood pressure and anthropometric measurements of all individuals who participated in the study and retrospective 24-hour food consumption records were recorded again and the study was concluded.
  Other Names: hypocaloric diet intervention; weight loss intervention
  Arms: Intervention Group

SUMMARY:
This study evaluated the effects of a weight loss diet on biochemical, anthropometric variables, and cluster of differentiation 36 (CD36) levels in 65 patients newly diagnosed with metabolic syndrome (MetS). Participants followed an 8-week medical nutrition therapy (MNT) designed to achieve at least 5% weight loss. Significant changes were observed in some biochemical parameters and blood pressure among those who adhered to the diet. CD36 levels showed correlations with various metabolic and body composition parameters.

DETAILED DESCRIPTION:
This research aimed to assess the impact of a weight loss diet on biochemical and anthropometric variables, as well as CD36 levels, in 80 patients newly diagnosed with metabolic syndrome (MetS) who began a weight loss program. The study was completed all of whom were diagnosed with MetS and had applied to the Internal Medicine Outpatient Clinic at Ordu University Training and Research Hospital. At the start of the study, participants were provided with medical nutrition therapy (MNT) tailored to their energy and nutritional needs, as well as their lifestyle, with the goal of achieving at least a 5% weight loss within 8 weeks. Patients were monitored regularly throughout the process.

Before initiating MNT, participants' general characteristics and dietary habits were collected through face-to-face interviews. Additionally, 24-hour dietary recalls and anthropometric measurements were taken both before and at the end of the 8th week. Biochemical data were retrieved from patient records, blood pressure was measured by a physician, and fasting blood samples were collected for CD36 analysis, which were then stored at -80°C until further examination.

By the end of the study, some individuals adhered strictly to the MNT. Statistical differences were observed in some biochemical parameters and blood pressure between those who complied with MNT and those who did not. Correlations were observed between CD36 levels and some variables.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 19-64
* Being diagnosed with MetS by a physician according to the International Diabetes Federation (IDF)-2005 metabolic syndrome diagnostic criteria
* Being a volunteer to participate in the study

Exclusion Criteria:

* Being pregnant and breastfeeding
* Smoking and drinking alcohol
* Having any chronic disease other than metabolic syndrome
* Taking regular medication
* Taking regular nutritional supplements
* Having a change in weight within the last 3 months

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Change in the intervention group | Week 0 - Week 8
  A decrease in body weight, improvement in biochemical findings and a decrease in serum CD36 levels are expected in individuals who follow the given diet.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet FISUNOGLU, Assoc. Prof., Study Director — Hacettepe University; Ozlem Ozdemir, Assist. Prof, Study Chair — Ordu University
Locations (1):
- Ordu University, Ordu, Altınordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I do not want to share this before publishing the research as a research article.

REFERENCES:
- [Result] Khaleel AA, Al-Barzinji RMGT. Soluble CD36 Concentration in Diabetic Hypertensive Patients with Coronary Atherosclerosis. Cell Mol Biol (Noisy-le-grand). 2022 May 22;68(1):109-116. doi: 10.14715/cmb/2022.68.1.14. PMID 35809322
- [Result] Rac ME, Safranow K, Garanty-Bogacka B, Dziedziejko V, Kurzawski G, Goschorska M, Kuligowska A, Pauli N, Chlubek D. CD36 gene polymorphism and plasma sCD36 as the risk factor in higher cholesterolemia. Arch Pediatr. 2018 Apr;25(3):177-181. doi: 10.1016/j.arcped.2018.01.008. Epub 2018 Mar 23. PMID 29576254
- [Result] Blomquist C, Chorell E, Ryberg M, Mellberg C, Worrsjo E, Makoveichuk E, Larsson C, Lindahl B, Olivecrona G, Olsson T. Decreased lipogenesis-promoting factors in adipose tissue in postmenopausal women with overweight on a Paleolithic-type diet. Eur J Nutr. 2018 Dec;57(8):2877-2886. doi: 10.1007/s00394-017-1558-0. Epub 2017 Oct 26. PMID 29075849
- [Result] do Amaral CL, Milagro FI, Curi R, Martinez JA. DNA methylation pattern in overweight women under an energy-restricted diet supplemented with fish oil. Biomed Res Int. 2014;2014:675021. doi: 10.1155/2014/675021. Epub 2014 Jan 22. PMID 24579084
- [Result] Mora-Rodriguez R, Ortega JF, Morales-Palomo F, Ramirez-Jimenez M. Weight loss but not gains in cardiorespiratory fitness after exercise-training predicts improved health risk factors in metabolic syndrome. Nutr Metab Cardiovasc Dis. 2018 Dec;28(12):1267-1274. doi: 10.1016/j.numecd.2018.08.004. Epub 2018 Aug 23. PMID 30459053
- [Result] Alkhatatbeh MJ, Ayoub NM, Mhaidat NM, Saadeh NA, Lincz LF. Soluble cluster of differentiation 36 concentrations are not associated with cardiovascular risk factors in middle-aged subjects. Biomed Rep. 2016 May;4(5):642-648. doi: 10.3892/br.2016.622. Epub 2016 Mar 3. PMID 27123261
- [Result] Yanai H, Chiba H, Morimoto M, Jamieson GA, Matsuno K. Type I CD36 deficiency in humans is not associated with insulin resistance syndrome. Thromb Haemost. 2000 May;83(5):786. No abstract available. PMID 10823279
- [Result] Furuhashi M, Ura N, Nakata T, Shimamoto K. Insulin sensitivity and lipid metabolism in human CD36 deficiency. Diabetes Care. 2003 Feb;26(2):471-4. doi: 10.2337/diacare.26.2.471. PMID 12547883
- [Result] Lopez-Carmona MD, Plaza-Seron MC, Vargas-Candela A, Tinahones FJ, Gomez-Huelgas R, Bernal-Lopez MR. CD36 overexpression: a possible etiopathogenic mechanism of atherosclerosis in patients with prediabetes and diabetes. Diabetol Metab Syndr. 2017 Jul 18;9:55. doi: 10.1186/s13098-017-0253-x. eCollection 2017. PMID 28729885
- [Result] Griffin E, Re A, Hamel N, Fu C, Bush H, McCaffrey T, Asch AS. A link between diabetes and atherosclerosis: Glucose regulates expression of CD36 at the level of translation. Nat Med. 2001 Jul;7(7):840-6. doi: 10.1038/89969. PMID 11433350
- [Result] Marechal L, Laviolette M, Rodrigue-Way A, Sow B, Brochu M, Caron V, Tremblay A. The CD36-PPARgamma Pathway in Metabolic Disorders. Int J Mol Sci. 2018 May 21;19(5):1529. doi: 10.3390/ijms19051529. PMID 29883404
- [Result] Pardina E, Ferrer R, Rossell J, Ricart-Jane D, Mendez-Lara KA, Baena-Fustegueras JA, Lecube A, Julve J, Peinado-Onsurbe J. Hepatic CD36 downregulation parallels steatosis improvement in morbidly obese undergoing bariatric surgery. Int J Obes (Lond). 2017 Sep;41(9):1388-1393. doi: 10.1038/ijo.2017.115. Epub 2017 May 10. PMID 28555086
- [Result] Botha J, Nielsen MH, Christensen MH, Vestergaard H, Handberg A. Bariatric surgery reduces CD36-bearing microvesicles of endothelial and monocyte origin. Nutr Metab (Lond). 2018 Oct 23;15:76. doi: 10.1186/s12986-018-0309-4. eCollection 2018. PMID 30386406
- [Result] Knosgaard L, Kazankov K, Birkebaek NH, Holland-Fischer P, Lange A, Solvig J, Horlyck A, Kristensen K, Rittig S, Vilstrup H, Gronbaek H, Handberg A. Reduced sCD36 following weight loss corresponds to improved insulin sensitivity, dyslipidemia and liver fat in obese children. Eur J Clin Nutr. 2016 Sep;70(9):1073-7. doi: 10.1038/ejcn.2016.88. Epub 2016 Jun 8. PMID 27273071